CLINICAL TRIAL: NCT04955093
Title: An Investigation Into the Use of Heart Rate Variability Biofeedback in People With Autistic Spectrum Disorder
Brief Title: Heart Rate Variability Biofeedback in Young People With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: South Eastern Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRAS139122; 15/NI/0255 (Other: UK-HRA-REC)
Record Dates: First submitted 2017-09-19; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Autistic Disorders Spectrum
MeSH Terms: conditions — Child Development Disorders, Pervasive | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Feasibility study to test out methodology prior to any future large scale trial.
  It involves a detailed follow up of a clinical sample of people with highfunctioning autism, using repeated measures in a randomized control experimental design. Intervention participants will be given a biofeedback device and training immediately, whilst the control group will wait 6 weeks and then receive the intervention. This will help to increase participation and maximize the detailed data collection that is required
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Device: Biofeedback
- Control (No Intervention)

INTERVENTIONS:
Device: Biofeedback — Technology to provide Heart Rate Variability Biofeedback
  Arms: Intervention

SUMMARY:
Biofeedback is a process that allows people to obtain information about their internal physiological reactions and thereby learn to control them.

Researchers studying the brain and nervous system have found that regulating heart rate can help us to relax. Controlling heart rate using biofeedback has been shown in some studies to help people manage symptoms of stress such as anxiety and depression.

This research will explore whether biofeedback can help people with autism or Asperger syndrome reduce reported symptoms of stress.

Participants with a diagnosis of high functioning autism will be invited to use a biofeedback device that helps them to regulate their heart rate. People who enrol for the study will be randomly assigned different biofeedback devices. Training and support in the use of the device will be provided to participants.

Assessment will involve obtaining questionnaire reports from participants and their carers about participant levels of anxiety, depression and sensory symptoms, demographics and lifestyle. These assessments will be carried out at the beginning, in the middle and at the end of the study to see if there are any differences in how each participant's heart rate changes, whether there are any changes in participant's reported symptoms. Participants will be asked to give daily reports on their progress to monitor stress levels, usability of device and dropout rates. The overall aim is to determine whether biofeedback is a way of helping people with autism to reduce symptoms of stress.

DETAILED DESCRIPTION:
Based on a review of the literature, it is hypothesised that HRV biofeedback could offer a means to help regulate ANS dysfunction and symptoms such as anxiety & depression in people with autistic spectrum disorder. To date, no studies have been identified which report on the pre post measurement of HRV in autism using a longitudinal design. Furthermore, to date, no published studies have reported on the use of portable HRV biofeedback devices as a potential intervention for individuals with autism to help manage symptoms such as anxiety & depression.

An initial usability evaluation has been carried out and approved by Ulster University faculty of Life & Health sciences in 2014 to determine the timings required to undertake the assessment and assess usability of equipment, measures, physiological assessment sensors and recording of data (see appendix I for a summary). The current study aims to assess the feasibility of employing a technology intervention for people with autism using small portable HRV biofeedback devices to help manage symptoms such as anxiety. Because of the differences in physiology seen in many people with autism, any study aiming to understand a potential new intervention for this population should include pre and post intervention assessments of they react physiologically and respond to information. This study will therefore use pre and post questionnaire assessment from participants and their carers, but will also record participant's heart rate variability pre and post intervention to assess any changes in participants underlying physiology.

Aim To understand the use of heart rate variability biofeedback in people with autistic spectrum disorder.

Objectives

1. To provide a home based HRV biofeedback intervention to people with autistic spectrum disorder.
2. To collect data from participants and their carers on participant anxiety, depression and physiological arousal before and after using a biofeedback device.
3. To assess the adoption of HRV biofeedback technology in terms of user acceptance and levels of dropout.
4. To evaluate the risks and benefits of this technology in terms of stress management.
5. To develop recommendations on the use of HRV biofeedback for people with autistic spectrum disorder.

Methodology The study will follow the revised MRC guidelines for the development and evaluation of complex interventions, namely a feasibility and piloting study which will look at dropout rates, test methodology and procedure, and determine the size of sample that would eventually be needed to obtain estimates of effect size in a full scale randomised trial.

Design The study is essentially a clinical trial that involves a detailed follow up of a sample of people with autistic spectrum disorder (n=39, IQ>70) using repeated measures in a randomised control experimental design.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of High functioning autism / Asperger's syndrome using standardized tests (ADOS / ADI / DISCO), IQ over 70, English speaker Existing or previous client resident within South Eastern Health & Social Care Trust catchment area.

Exclusion Criteria:

Learning disability (IQ<70). Cardiac condition / pacemaker. Drug /alcohol addiction Current psychosis Current suicidal ideation. Eczema / psoriasis Immunosuppressing condition MRSA / C Difficile

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Reduction in Anxiety Scale using Beck Youth Inventory | At baseline, after six weeks and at end-point at 12 weeks
  10-15 minute Questionnaire

SECONDARY OUTCOMES:
Any change in Heart rate variability (ideally key metrics increased) | At baseline, after six weeks and at end-point at 12 weeks
  Physiological recording of heart rate variability using single lead ECG

CONTACTS AND LOCATIONS:
Locations (1):
- South Eastern Health Trust, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Coulter H, Donnelly M, Mallett J, Kernohan WG. Heart Rate Variability Biofeedback to Treat Anxiety in Young People With Autism Spectrum Disorder: Findings From a Home-Based Pilot Study. JMIR Form Res. 2022 Aug 26;6(8):e37994. doi: 10.2196/37994. PMID 36018712